CLINICAL TRIAL: NCT01426581
Title: Effectiveness of Interventions to Teach Respiratory Inhaler techNique (E-TRaIN)
Acronym: E-TRaIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 11-0248
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-10

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Asthma; Chronic Obstructive Pulmonary Disease (COPD); Pulmonary Disease, Chronic Obstructive; Lung Disease, Obstructive; Self-management; Health Literacy
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational Intervention A (Experimental): Intervention: Teach to Goal
  Interventions: Behavioral: Teach-To-Goal
- Educational Intervention B: (Experimental): Brief Intervention
  Interventions: Behavioral: Brief Intervention

INTERVENTIONS:
Behavioral: Teach-To-Goal — Participants observe a demonstration on the use of each inhaler, with corresponding verbal step-by-step instructions (demonstration, verbal instruction), then participants 'teachback" or re-demonstrate the steps; cycles are repeated are read step-by-step instructions (verbal instructions) for each respective inhaler (Metered Dose Inhaler +/- Diskus), and receive a copy of these instructions with images depicting the steps (written instructions)
  Arms: Educational Intervention A
Behavioral: Brief Intervention — Participants are read step-by-step instructions (verbal instructions) for each respective inhaler (Metered Dose Inhaler +/- Diskus), and receive a copy of these instructions with images depicting the steps (written instructions)
  Arms: Educational Intervention B:

SUMMARY:
The purpose of this study is to evaluate the relative effectiveness of two different ways to teach subjects while hospitalized how to use respiratory inhalers and to follow-up after discharge home from the hospital to determine durability of the education.

Teach-to-Goal (TTG) education employs instruction followed by patient "teach-back," then repeated cycles of learning and assessment until a skill is mastered. By contrast, Brief Intervention (BI) education only consists of providing the patient with verbal and written instruction.

The investigators hypothesize that hospital-based TTG compared to BI increases a patient's ability to retain instructions on respiratory inhaler technique. The investigators will test this hypothesis separately for the MDI and Diskus® devices after discharge.

DETAILED DESCRIPTION:
Respiratory inhalers are often used incorrectly by patients with obstructive lung disorders (including patients hospitalized with exacerbations of asthma or chronic obstructive pulmonary disease (COPD). As the mainstay of bronchodilator and anti-inflammatory therapy in patients with OLD, the implication of this difficulty with self-management is that patients are at risk for under-treatment and worse health outcomes. Several factors are thought to contribute to poor self-management skills, particularly inadequate patient education at healthcare encounters and inadequate patient health literacy. However, the most effective strategy to instruct patients about respiratory inhaler use in hospital settings is unclear, particularly in populations enriched with inadequate health literacy.

Therefore, the overall goal of this study is to evaluate the relative effectiveness of two hospital-based educational interventions: Teach-To-Goal (TTG, iterative cycles of demonstration-based education and assessment) versus Brief Intervention (BI, one-time set of verbal instructions) on the durability of instructions provided in the hospital and its effect on clinical outcomes (e.g., respiratory events and/or death), post hospital discharge. The investigators also plan to evaluate whether the relative effectiveness of TTG vs. BI varies by level of health literacy. The objectives of this proposal are to conduct a study in adults hospitalized with asthma/COPD to 1) to evaluate the relative effectiveness of hospital-based TTG versus BI on patients' ability to retain instruction about the correct use of MDI and Diskus® devices after discharge home and 2) To determine the relative effectiveness of TTG compared to BI for patients with less-than-adequate health literacy compared to those with adequate health literacy. These data will inform the development of a larger, multi-center clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Admitting diagnosis of asthma or COPD
* Physician- diagnosed asthma, asthma/COPD, or COPD. We will enroll patients even if the primary reason for admission is not asthma or COPD (e.g., patients admitted for heart failure, but with a physician diagnosis of COPD are eligible)
* Patient will be discharged home on a Metered Dose Inhaler (MDI; e.g., albuterol)

Exclusion Criteria:

* Currently in an intensive care unit
* Physician declines to provide consent
* Patient unable to provide consent (e.g., history of cognitive impairment, unable to understand English) or declines to provide consent
* Previous participant in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie G Press, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Press VG, Arora VM, Trela KC, Adhikari R, Zadravecz FJ, Liao C, Naureckas E, White SR, Meltzer DO, Krishnan JA. Effectiveness of Interventions to Teach Metered-Dose and Diskus Inhaler Techniques. A Randomized Trial. Ann Am Thorac Soc. 2016 Jun;13(6):816-24. doi: 10.1513/AnnalsATS.201509-603OC. PMID 26998961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized into TTG or BI between September 2011 and February 2013. Of the 120 participants, 100 were enrolled at hospital #1 and 20 were enrolled from hospital #2.
Groups:
- Teach To Goal: Intervention: Teach to Goal
  Teach-To-Goal: Participants observe a demonstration on the use of each inhaler, with corresponding verbal step-by-step instructions (demonstration, verbal instruction), then participants 'teachback" or re-demonstrate the steps; cycles are repeated are read step-by-step instructions (verbal instructions) for each respective inhaler (Metered Dose Inhaler +/- Diskus), and receive a copy of these instructions with images depicting the steps (written instructions)
- Brief Intervention:: Brief Intervention
  Brief Intervention: Participants are read step-by-step instructions (verbal instructions) for each respective inhaler (Metered Dose Inhaler +/- Diskus), and receive a copy of these instructions with images depicting the steps (written instructions)
Period: Overall Study
Arm/Group | Teach To Goal | Brief Intervention:
Started | 62 | 58
Completed | 62 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Brief Intervention: Brief Intervention
  Brief Intervention: Participants are read step-by-step instructions (verbal instructions) for each respective inhaler (Metered Dose Inhaler +/- Diskus), and receive a copy of these instructions with images depicting the steps (written instructions)
- Total: Total of all reporting groups
Arm/Group | Teach To Goal | Brief Intervention | Total
Number analyzed (Participants) | 62 | 58 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 51 | 105
  >=65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 88
  Male | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With MDI Misuse From Baseline to 30 Days Post-Discharge
Description: To evaluate the relative effectiveness of hospital-based TTG versus BI on patients' ability to retain instruction about the correct use of MDI Devices one month after discharge home.
Time Frame: 1 month
Measure: Number; unit: percentage
Groups:
- Teach to Goal: Teach-To-Goal: Participants observe a demonstration on the use of each inhaler, with corresponding verbal step-by-step instructions (demonstration, verbal instruction), then participants 'teachback" or re-demonstrate the steps; cycles are repeated are read step-by-step instructions (verbal instructions) for each respective inhaler (Metered Dose Inhaler +/- Diskus), and receive a copy of these instructions with images depicting the steps (written instructions)
Arm/Group | Teach to Goal | Brief Intervention
Number analyzed (Participants) | 62 | 58
percentage
  Misuse at Baseline | 92 | 84
  Misuse at 30 days post-discharge | 11 | 60

2. Secondary Outcome: Role of Health Literacy - Number of Less-Than-Adequate Health Literacy Participants With 30 Days Post Discharge Acute-Care Events
Description: To determine the relative effectiveness of TTG compared to BI for patients with less-than-adequate health literacy using self-reported acute-care events 30 days post discharge. To measure less-than-adequate health literacy, the investigators administered the Short Test of Functional Health Literacy in Adults, a validated tool to assess whether a participant has adequate, marginal, or inadequate health literacy. Less-than-adequate included marginal and inadequate health literacy.
Time Frame: 1 month
Population: Out of 120 participants, 23 were screened to have less-than-adequate health literacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Teach To Goal | Brief Intervention
Number analyzed (Participants) | 13 | 10
Participants | 2 | 7

3. Secondary Outcome: Number of Participants With Self-Efficacy
Description: This is a self-reported measure of how confident a participant is on how well they use their metered dose inhaler.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Teach To Goal | Brief Intervention:
Number analyzed (Participants) | 62 | 58
Participants | 49 | 38

4. Secondary Outcome: Symptom Control
Description: Symptom control will be assessed using interviewer-administered surveys. Using the Borg Dyspnea Scale, a validated Scale from 0 - 20 where 20 is maximal dyspnea, we took the difference between the the 30 day follow-up self reported shortness of breath from baseline to see if there was improvement in symptom control.
Time Frame: 1 month
Population: The discrepancy from the number of participants in each group and the number of participants analyzed is due to missing data values due to lose to follow-up for the 30-day post discharge visit. 8 participants did not have values in the Teach To Goal group and 5 did not for the Brief Intervention group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teach To Goal | Brief Intervention:
Number analyzed (Participants) | 54 | 53
units on a scale | -1.69 (2.75) | -1.43 (2.59)

5. Secondary Outcome: Number of Participants With Acute Care Events 30 Days Post Discharge
Description: Exacerbation/acute care events within one month of hospital discharge
Time Frame: 1 month
Population: The discrepancy between the number of participants analyzed in each group and the number of participants in each arm total is due to lost to follow-up. In the Teach to Goal arm, 8 participants were lost to follow up and 5 participants were lost to follow up in the Brief Intervention arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Teach To Goal | Brief Intervention:
Number analyzed (Participants) | 54 | 53
Participants | 9 | 19

ADVERSE EVENTS:
Arm/Group | Educational Intervention A | Educational Intervention B:
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/58
Other Adverse Events (participants affected / at risk) | 0/62 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No